CLINICAL TRIAL: NCT06123182
Title: Guided Episodic Future Thinking to Increase Physical Activity Adherence and Promote Healthy Brain Aging Among Mid-Life Adults: Phase II
Brief Title: Guided Episodic Future Thinking to Increase Physical Activity Adherence and Promote Healthy Brain Aging
Acronym: GETActiveHIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Laura Martin, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00150353; R33AG078087 (NIH)
Record Dates: First submitted 2023-10-27; First posted 2023-11-08 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Exercise Training; Aging
Keywords: Adherence; Guided Imagery

STUDY DESIGN:
Intervention Model Description: 2 (positive affect imagery vs. neutral) x 2 (episodic future thinking vs. recent thinking)
Who Masked: Participant, Investigator
Masking Description: Primary investigator is masked to intervention assignment. Participants are masked to the intervention - however may be able to figure out intervention based on the guided imagery content
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Episodic Future Thinking (EFT) + Positive Affective Imagery (PAI) (Experimental): Assigned guided imagery will be delivered during each exercise session throughout the 6-week exercise program. The guided imagery recordings will be delivered via audio recording during warm-up and cool-down periods during in-lab exercise sessions. The EFT will always be delivered during warm-up and the PAI will always be delivered during cool-down.
  Interventions: Behavioral: Episodic Future Thinking; Behavioral: Positive Affective Imagery; Behavioral: HIIT Exercise Intervention
- Episodic Future Thinking (EFT) + Neutral Affective Imagery (NAI) (Experimental): Assigned guided imagery will be delivered during each exercise session throughout the 6-week exercise program. The guided imagery recordings will be delivered via audio recording during warm-up and cool-down periods during in-lab exercise sessions. The EFT will always be delivered during warm-up and the NAI will always be delivered during cool-down.
  Interventions: Behavioral: Episodic Future Thinking; Behavioral: Neutral Affective Imagery; Behavioral: HIIT Exercise Intervention
- Episodic Recent Thinking (ERT) + Positive Affective Imagery (PAI) (Experimental): Assigned guided imagery will be delivered during each exercise session throughout the 6-week exercise program. The guided imagery recordings will be delivered via audio recording during warm-up and cool-down periods during in-lab exercise sessions. The ERT will always be delivered during warm-up and the PAI will always be delivered during cool-down.
  Interventions: Behavioral: Episodic Recent Thinking; Behavioral: Positive Affective Imagery; Behavioral: HIIT Exercise Intervention
- Episodic Recent Thinking (ERT) + Neutral Affective Imagery (NAI) (Active Comparator): Assigned guided imagery will be delivered during each exercise session throughout the 6-week exercise program. The guided imagery recordings will be delivered via audio recording during warm-up and cool-down periods during in-lab exercise sessions. The ERT will always be delivered during warm-up and the NAI will always be delivered during cool-down.
  Interventions: Behavioral: Episodic Recent Thinking; Behavioral: Neutral Affective Imagery; Behavioral: HIIT Exercise Intervention

INTERVENTIONS:
Behavioral: Episodic Future Thinking — During the audio recorded guided imagery exercise participants will be asked to think in detail of a future (6 months to a year) where they have made healthy choices regarding physical activity and are physically active.
  Arms: Episodic Future Thinking (EFT) + Neutral Affective Imagery (NAI); Episodic Future Thinking (EFT) + Positive Affective Imagery (PAI)
Behavioral: Episodic Recent Thinking — During the audio recorded guided imagery exercise participants will be asked to think about a routine weekly activity.
  Arms: Episodic Recent Thinking (ERT) + Neutral Affective Imagery (NAI); Episodic Recent Thinking (ERT) + Positive Affective Imagery (PAI)
Behavioral: Positive Affective Imagery — During the audio recorded guided imagery exercise participants will be asked to think in detail about the positive outcomes and sensations associated with an exercise bout.
  Arms: Episodic Future Thinking (EFT) + Positive Affective Imagery (PAI); Episodic Recent Thinking (ERT) + Positive Affective Imagery (PAI)
Behavioral: Neutral Affective Imagery — During the audio recorded guided imagery exercise participants will be asked to think in detail about the physical sensations associated with an exercise bout.
  Arms: Episodic Future Thinking (EFT) + Neutral Affective Imagery (NAI); Episodic Recent Thinking (ERT) + Neutral Affective Imagery (NAI)
Behavioral: HIIT Exercise Intervention — The high intensity interval training (HIIT) will be conducted 2 times per week for 6 weeks. The duration of each individual exercise session will last about 45 minutes. After the 5-minute warm-up at 30% peak workload, HIIT will consist of repeated 1-minute high intensity bursts ("on" interval) alternated with 1-minute interval recovery ("off" interval) for 25 minutes. The "on" interval will begin at 80% of peak watts (range: 75%-85%) followed by the "off" interval at 10% of peak watts. The session will end with up to 10 minute cool-down at 20% peak workload.

SUMMARY:
The goal of this behavioral clinical trial is to learn how to increase physical activity in mid-life adults. Specifically, can guided imagery that includes creating mental pictures increase excitement about working out.

Participants will be asked to complete testing at the beginning of the study, following 6-weeks of an in-person exercise program, and 6-weeks after finishing the exercise program. Testing will include an exercise test, MRI, questionnaires, computer tasks, and a blood draw.

DETAILED DESCRIPTION:
The proposed project will target regulation and reward systems using guided imagery to increase exercise adherence by increasing positive affect and the evaluation of future rewards among mid-life adults. The investigators will conduct a within subject design in 160 mid-life adults (45-65 years of age) and examine the impact of different components of guided imagery on exercise adherence, regulation systems indexed by delay discounting, positive affect related to exercise, and functional neuroimaging (i.e., connectivity between regulation and reward brain regions). Participants will be asked to complete three assessment appointment periods: 1) baseline, 2) 6-weeks (i.e., end of exercise intervention), and 3) 12-weeks. Each appointment will include assessment of primary outcome measures of delay discounting and exercise positive affect. In addition, baseline and 6-week appointments will include functional magnetic resonance imaging (fMRI) assessments of functional connectivity between reward and regulation regions. Physical activity will be measured at baseline, immediately following the intervention, and 6 weeks following the intervention to explore changes in physical activity across study participation. At the end of the final appointment participants will be debriefed on the goals of the study and asked to provide feedback related to feasibility, the guided imagery experience, and exercise intervention experience to inform future research. In addition, blood draws will be completed at baseline to assess genetic risk for developing Alzheimer's disease (i.e., APOE). If successful, this approach could be used in future studies to increase participation in exercise and adherence to exercise interventions with the goal of promoting brain health and reducing the risk of developing Alzheimer's disease. The design of the proposed clinical trial permits a rigorous evaluation of the role of engaging regulation and reward systems to change immediate and future reward. The exercise intervention will consist of one-on-one high intensity interval training (HIIT) overseen by an exercise specialist twice a week for 6 weeks. Exercise adherence will be monitored as the percentage of the weekly exercise and adherence to the HIIT protocol.

ELIGIBILITY:
Inclusion Criteria:

* speak English
* have access to reliable communication (a telephone or cell phone, computer, etc.)
* normal or corrected to normal vision and hearing
* ambulatory (without the use of assistive devices)
* physically underactive
* able to give informed consent
* able to exercise continuously on the recumbent stepper exercise device for 4 minutes greater than or equal to 25 watts to demonstrate ability to perform exercise on stepper & no aerobic exercise contraindications or other safety/physical concerns
* able to communicate with investigators, follow 2-step command & correctly answer consent comprehension questions
* stable blood pressure and statin medication doses for 30 days as these affect vascular health/hemodynamics
* willing and able to safely enter magnetic resonance (MR) scanner and attempt the MR scan
* willing and able to attempt a blood draw

Exclusion Criteria:

* patients with arrhythmias or acute cardiac events will be excluded due to potential complications with the supervised moderate exercise
* at risk for hazard due to magnetic fields due to MR safety concerns
* have any neurologic or psychiatric disorder except depression, anxiety (including post-traumatic stress disorder)
* have history of seizures or head trauma due to MR data quality

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Adherence to HIIT exercise | 1 to 6-weeks
  Adherence will be calculated as percent sessions attended each week and percent minutes during which the participant adhered to the HIIT protocol.
The Monetary-Choice Questionnaire | 1 to 6-weeks
  The Monetary-Choice Questionnaire is a 27-item self-administered questionnaire. For each item, the participant chooses between a smaller, immediate monetary reward and a larger, delayed monetary reward. The investigators will behaviorally assess participants' preferences for immediately available smaller rewards vs. delayed larger rewards.
Positive Affect | 1 to 6-weeks
  The Feeling Scale is a single item measure of core affect on which participants are asked to rate their current feelings on an 11-point scale ranging from -5 (very bad) to 5 (very good).

SECONDARY OUTCOMES:
Percent signal change in Functional Connectivity Neuroimaging | 1 to 6-weeks
  The investigators will assess % signal changes in brain connectivity between reward and regulation brain regions following intervention.

OTHER OUTCOMES:
Number of Participants with Alzheimer's Disease Risk | Baseline
  Genetic risk for Alzheimer's disease will be measured by examining APOE4 carrier status.
The Monetary-Choice Questionnaire | 1 to 12 weeks
  The Monetary-Choice Questionnaire is a 27-item self-administered questionnaire. For each item, the participant chooses between a smaller, immediate monetary reward and a larger, delayed monetary reward. The investigators will behaviorally assess participants' preferences for immediately available smaller rewards vs. delayed larger rewards.
Positive Affect | 1 to 12 weeks
  The Feeling Scale is a single item measure of core affect on which participants are asked to rate their current feelings on an 11-point scale ranging from -5 (very bad) to 5 (very good).
Amount of Daily Moderate to Vigorous Physical Activity (MVPA minutes) | 1 to 12 weeks
  The investigators will measure physical activity (MVPA minutes) at baseline, end of intervention, and end of follow-up using accelerometers worn daily for 10-14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Martin, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States